CLINICAL TRIAL: NCT03114618
Title: Genomic Predictors Indicating the Risk of Venous Thromboembolic Disease in Cancer Patients Treated in Outpatient Clinics
Brief Title: A New Clinic-Genetic Risk Score for Predicting Venous Thromboembolic Events in Cancer Patient
Acronym: ONCOTHROMB
Status: Completed | Type: Observational
Sponsor: Andres muñoz (Other)
Collaborators: Servicio de Oncología Médica. HGU Gregorio Marañón. Madrid (Unknown); Unitat de Genòmica de Malalties Complexes. Institut d'Investigació Sant Pau (Unknown); Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario de Fuenlabrada (Other); Hospital Universitario Marqués de Valdecilla (Other); Complexo Hospitalario de Ourense (Other); Complejo Universitario Torrecárdenas, Almería (Unknown); Gendiag (Industry); Ferrer inCode, S.L. (Industry); Unitat d'Hemostasia i Trombosi. Hospital de la Santa Creu i Sant Pau (Unknown); LEO Pharma (Industry); Sociedad Española de Trombosis y Hemostasia (SETH) (Unknown); Sociedad Española de Oncología Médica (SEOM) (Unknown); University Hospital Virgen de las Nieves (Other); Hospital Obispo Polanco, Teruel (Unknown); Complejo Hospitalario Universitario de Vigo (Other); Hospital General Universitario Elche (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Hospital General de Ciudad Real (Other)
Responsible Party: Sponsor-Investigator, Andres muñoz, MD PhD, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: ONCOTHROMB12-01
Record Dates: First submitted 2017-03-14; First posted 2017-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cancer-associated Thrombosis; Genetic Predisposition
Keywords: Venous thrombosis; Cancer; Risk Model Assessment; Genomic
MeSH Terms: conditions — Genetic Predisposition to Disease; Venous Thrombosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Venous thromboembolism (VTE) is a common disease in cancer patients and one of the major causes of cancer-associated mortality. Risk for developing VTE increases when cancer patients are receiving chemotherapy. Current risk scores for predicting cancer-associated VTE in ambulatory patients had low/moderate discrimination and clinical sensitivity. These models use clinical and biochemical parameters of the patient.

In the development of VTE genetics play a relevant role. The product Thrombo inCode (TiC) assess VTE risk prediction by using a combination of a genetic risk score (GRS) and clinical parameters from the patient. The investigators hypothesized that the GRS included in TiC combined with clinical parameter some of them associated with cancer could be better predicted by TiC than by current risk scores (Khorana score).

After publishing the primary results in 2018, we have expanded the GRS in a external validation cohort adding gliomas and biliary tract tumors. Also we have incorporated the assessment of D-dimer in order to improve the predictive capability.

DETAILED DESCRIPTION:
The working hypothesis of this study establishes that the risk of cancer patients suffering a thromboembolic event is conditioned by individual genomic factors. The genes to be analyzed have clearly demonstrated their relationship with thromboembolic disease in other clinical contexts. This study is considered the initiation of a field of research in genomic risk markers indicating a risk of thrombosis in cancer patients. The ultimate goal of the study is to establish a clinic-genomic score for selecting patients with a high risk of suffering thrombotic events who can benefit from guided thromboprophylaxis. Its secondary goal is to prevent the adverse effects of ineffective therapies in other patients (low-risk patients not requiring an anti-thrombotic prophylaxis).

The aim is to demonstrate the link between the clinic-genetic profile and the risk of suffering thromboembolic events in the group of cancer patients. The working hypothesis establishes that cancer patients who develop thrombotic events will have a higher score for the thrombosis risk clinic-genetic profile than cancer patients not developing thromboembolic events. The second aim is to analyze whether the thrombosis clinic-genetic risk score improves the detection of patients at risk of suffering a thromboembolic event compared to the Khorana predictive model routinely used (Khorana score).

Current validations ongoing:

An external retrospective validation adding 250 patients more and including D-dimer and other types of high-risk neoplasm.

An external prospective validation (second ONCOTRHROMB12-01 cohort 2) adding 450 patients more and including D-dimer and other types of high-risk neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients treated in outpatient clinics with a documented histological or cytological diagnosis for non-microcytic lung, colorectal, biliary tract cancer, pancreatic or esophago-gastric cancer at an advanced stage, locally advanced or localized not previously treated with systemic chemotherapy and/or radiation therapy who are candidate for chemotherapy in outpatient setting.
* Performance status 0-2.
* Patients signing the study informed consent form.

Exclusion Criteria:

* Life expectancy of less than 3 months.
* Patients undergoing anti-coagulant treatment before the cancer diagnosis for reasons other than a concurrent venous thromboembolic event.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients diagnosed with colorectal, esophago-gastric, biliary tract, pancreas or lung cancer who have not previously been treated with chemotherapy or chemotherapy and radiation therapy and are candidate for chemotherapy in outpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2013-03; Primary Completion 2020-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism events | During the 18 months of follow up
  The development of venous thromboembolism will be registered

CONTACTS AND LOCATIONS:
Overall Officials: Andrés J. Muñoz Martín, MD PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (9):
- Spain (9):
  - Complejo Hospitalario Torrecárdenas, Almería, Almería
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Clinic, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Hospitalario de Orense, Ourense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Soria JM, Morange PE, Vila J, Souto JC, Moyano M, Tregouet DA, Mateo J, Saut N, Salas E, Elosua R. Multilocus genetic risk scores for venous thromboembolism risk assessment. J Am Heart Assoc. 2014 Oct 23;3(5):e001060. doi: 10.1161/JAHA.114.001060. PMID 25341889
- [Result] Rubio-Terres C, Soria JM, Morange PE, Souto JC, Suchon P, Mateo J, Saut N, Rubio-Rodriguez D, Sala J, Gracia A, Pich S, Salas E. Economic analysis of thrombo inCode, a clinical-genetic function for assessing the risk of venous thromboembolism. Appl Health Econ Health Policy. 2015 Apr;13(2):233-42. doi: 10.1007/s40258-015-0153-x. PMID 25652150
- [Result] Munoz Martin AJ, Ortega I, Font C, Pachon V, Castellon V, Martinez-Marin V, Salgado M, Martinez E, Calzas J, Ruperez A, Souto JC, Martin M, Salas E, Soria JM. Multivariable clinical-genetic risk model for predicting venous thromboembolic events in patients with cancer. Br J Cancer. 2018 Apr;118(8):1056-1061. doi: 10.1038/s41416-018-0027-8. Epub 2018 Mar 28. PMID 29588512
- [Derived] Munoz A, Ay C, Grilz E, Lopez S, Font C, Pachon V, Castellon V, Martinez-Marin V, Salgado M, Martinez E, Calzas J, Ortega L, Ruperez A, Salas E, Pabinger I, Soria JM. A Clinical-Genetic Risk Score for Predicting Cancer-Associated Venous Thromboembolism: A Development and Validation Study Involving Two Independent Prospective Cohorts. J Clin Oncol. 2023 Jun 1;41(16):2911-2925. doi: 10.1200/JCO.22.00255. Epub 2023 Feb 2. PMID 36730884